CLINICAL TRIAL: NCT03065062
Title: Phase I Study of the CDK4/6 Inhibitor Palbociclib (PD-0332991) in Combination With the PI3K/mTOR Inhibitor Gedatolisib (PF-05212384) for Patients With Advanced Squamous Cell Lung, Pancreatic, Head & Neck and Other Solid Tumors
Brief Title: Study of the CDK4/6 Inhibitor Palbociclib (PD-0332991) in Combination With the PI3K/mTOR Inhibitor Gedatolisib (PF-05212384) for Patients With Advanced Squamous Cell Lung, Pancreatic, Head & Neck and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Geoffrey Shapiro, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-499
Record Dates: First submitted 2017-02-06; First posted 2017-02-27 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer Squamous Cell; Solid Tumors; Head & Neck Cancer; Pancreatic Cancer
Keywords: Lung Cancer Squamous Cell; Head & Neck Cancer; Neoplasms; Endometrial Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Pancreatic Neoplasms; Neoplasms; Endometrial Neoplasms | interventions — palbociclib; gedatolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination Of Palbociclib and Gedatolisib (Experimental): * Palbociclib will be administered orally once daily on Days 1-21 for each of the 4-week cycles at a pre-determined dose.
  * Gedatolisib will be administered intravenously once weekly on the first day for each of the four weeks during the 4-week cycles at a pre-determined dose.
  Interventions: Drug: Palbociclib; Drug: Gedatolisib

INTERVENTIONS:
Drug: Palbociclib — Palbociclib will be administered orally once daily, 3 weeks out of every 4 in each cycle. The initial dose for part 1 of the study will be 100 mg daily. Dosing will be adjusted until Maximum Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D) are established. No pre-medications for palbociclib are required. It should be administered with food.
  Other Names: IBRANCE; PD-0332991
Drug: Gedatolisib — Gedatolisib will be administered once weekly on the first day for each of the four weeks during the 4-week cycle. The initial dose for part 1 of the study will be 110 mg. Dosing will be adjusted until Maximum Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D) are established. No pre-medications for gedatolisib are required.
  Other Names: PF-05212384

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for cancer that might have a specific change in the phosphatidylinositol-3 phosphate (PI3K) pathway.

DETAILED DESCRIPTION:
This research study is an open-label Phase I clinical trial, which tests the safety of an investigational drug or combination of investigational drugs and also tries to define the appropriate dose of the investigational drug(s) to use for further studies. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved Palbociclib for the participant specific disease but it has been approved for other uses. The FDA has not approved Gedatolisib alone or in combination with Palbociclb as a treatment option for the participant's disease.

In this research study the investigators hope to determine if treatment with Palbociclib and Gedatolisib will be tolerated and will help to shrink or stop the growth of the participant's cancer. Palbociclib is an oral drug which has been shown to stop the cell cycle, which is the way a cell initiates growth. Gedatolisib is thought to work by controlling a series of events directing cell growth and survival. Gedatolisib may work to stop or slow activity within tumor cells. By putting these two drugs together the investigators hope that it will have a greater effect on cancer growth than either drug alone.

ELIGIBILITY:
Inclusion Criteria:

* For Part I, participants must have histologically confirmed malignancy that is metastatic or unresectable and resistant to standard therapy or for which no standard therapy is available. For Part II, participants must have histologically confirmed advanced squamous cell lung cancer, advanced pancreatic cancer, advanced head & neck cancer (specifically non-oropharynx squamous cell carcinoma or HPV-negative oropharynx squamous cell carcinoma), or any tumor with suspected PI3K-pathway dependence (either by mutation or by known biologic rationale, such as endometrial cancer. PI3K dependence includes the presence of a PIK3CA-mutant hotspot mutation, PIK3CA copy number gain, or PTEN loss in the archival or fresh tumor tissue specimen identified in a CLIA-certified laboratory. All genetic findings must be reviewed by the study PI, prior to study entry.)
* For Part I, participants are required to have only evaluable disease (disease that is visible on imaging studies but does not meet RECIST criteria for measurable disease). For Part II, participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan. See section 10 for the evaluation of measureable disease.
* Participants are permitted to have any number of prior therapies prior to enrollment
* Age ≥ 18 years. .
* ECOG performance status ≤ 2
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Hemoglobin ≥9.0 gm/dL
  * Platelets ≥ 100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal (≤ 5.0 X institutional upper limit of normal permitted if hepatic metastases present)
  * Creatinine within 1.5x the ULN institutional limits
  * Fasting glucose ≤ 126 mg/dL (7.0 mmol/L)
  * HbA1c ≤ 7.0%
* The effects of palbociclib and Gedatolisib (PF-05212384) on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 90 days after discontinuation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from acute effects of any prior therapy to baseline or Grade ≤1 except for Alopecia or AEs not constituting a safety risk in the opinion of the investigator.
* Participants may not be receiving any other study agents concurrently with the study drugs.
* Participants with symptomatic brain metastases that require active treatment are excluded.
* Current use or anticipated need for food or medications that are known strong CYP3A4 inhibitors/inducers, including their administration within 7-days prior to the first Gedatolisib (PF-05212384) or palbocilib dose and during study treatment.
* QTc > 480 msec; history of QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes.
* Patients with a history of diabetes.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the study agents have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with the study agents, breastfeeding should be discontinued if the mother is treated.
* Individuals with a history of other malignancy are ineligible except for the following circumstances. Individuals with a history of previous malignancies are eligible if they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Active and clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Concurrent use or anticipated need for medications that are mainly metabolized by UGT1A9 including their administration within 7-days prior to the first dose of study drug.
* Current use or anticipated need for food or medications that are metabolized by CYP2D6, and of narrow therapeutic index including their administration within 10-days prior to the first Gedatolisib (PF-05212384) dose and during study treatment.
* Concurrent use of herbal preparations including saw palmetto.
* Current use of drugs known to prolong QT interval.
* Concurrent use of proton pump inhibitors (including, but not limited to, dexlansoprazole, esomeprazole, lansoprazole, omeprazole, pantoprazole, rabeprazole) with palbociclib is prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose and Recommended Phase 2 Dose | 2 years
  The dose-escalation schedule will use the mTPI design to discover the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of the combination of palbociclib and gedatolisib.
Incidence of Treatment-Emergent Adverse Events | 2 years
  Number of participants with treatment-related adverse events as assessed by version 4.0 of the NCI Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Progression Free Survival Rate at 4 months | 4 months
  Evaluate the preliminary clinical efficacy of palbociclib and gedatolisib in the following expansion cohorts: 1) advanced squamous cell lung cancer, 2) advanced pancreatic cancer, 3) advanced head & neck cancer, and 4) any tumor with presumed PI3K-pathway dependence using CT and MRI scans per RECIST version 1.
Target engagement of palbociclib and gedatolisib in paired tumor biopsies | 2 years
  Confirm target engagement of palbociclib and gedatolisib in pre- and on-treatment tumor biopsies from patients enrolled to the MTD expansion cohort through evaluation of changes in immunohistochemical staining for parameters of CDK and PI3K activity.
Pharmacokinetic parameter (maximum concentration [Cmax]) of gedatolisib in the absence or presence of palbociclib | At 0.5, 1, 2, 4, 6, 8, 10, 24, 72, 120 and 168 hours after dosing (lead-in dose 7 days prior to cycle 1 day 1, and cycle 1 day 15)
Pharmacokinetic parameter (area under the curve [AUC]) of gedatolisib in the absence or presence of palbociclib | At 0.5, 1, 2, 4, 6, 8, 10, 24, 72, 120 and 168 hours after dosing (lead-in dose 7 days prior to cycle 1 day 1, and cycle 1 day 15)
Pharmacokinetic parameter (half-life [t1/2]) of gedatolisib in the absence or presence of palbociclib | At 0.5, 1, 2, 4, 6, 8, 10, 24, 72, 120 and 168 hours after dosing (lead-in dose 7 days prior to cycle 1 day 1, and cycle 1 day 15)
Pharmacokinetic parameters (maximum concentration [Cmax]) of palbociclib in the presence of gedatolisib | At 1, 2, 4, 6, 8, 10, and 24 hours after dosing (cycle 1 day 15)
Pharmacokinetic parameters (area under the curve [AUC]) of palbociclib in the presence of gedatolisib | At 1, 2, 4, 6, 8, 10, and 24 hours after dosing (cycle 1 day 15)
Pharmacokinetic parameters (half-life [t1/2]) of palbociclib in the presence of gedatolisib | At 1, 2, 4, 6, 8, 10, and 24 hours after dosing (cycle 1 day 15)
Overall Response Rate | 2 years
  Evaluate the preliminary clinical efficacy of palbociclib and gedatolisib in advanced solid tumors using CT and MRI scans per RECIST version 1.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Shapiro, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No